CLINICAL TRIAL: NCT00489736
Title: Randomized Double Blind Trial to Evaluate the Efficacy and Safety of Dronedarone (400mg BID) Versus Amiodarone (600mg Daily for 28 Days, Then 200mg Daily Thereafter) for at Least 6 Months for the Maintenance of Sinus Rhythm in Patients With Atrial Fibrillation (AF)
Brief Title: Efficacy & Safety of Dronedarone Versus Amiodarone for the Maintenance of Sinus Rhythm in Patients With Atrial Fibrillation
Acronym: DIONYSOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: International Clinical Development, Clinical Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC4968
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Results first posted 2009-11-09 (Estimated); Last update posted 2010-02-18 (Estimated); Status verified 2010-02

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; sinus rhythm; amiodarone
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dronedarone; Amiodarone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dronedarone 400mg bid (Experimental): dronedarone 400mg tablets administered twice a day (bid) and matching over-encapsulated tablets of placebo of amiodarone 200mg
  Interventions: Drug: dronedarone (SR33589)
- Amiodarone 600mg/200mg od (Active Comparator): over-encapsulated tablets of amiodarone 200mg (600mg daily for 28 days then 200mg daily) administered once daily (od) and matching placebo of dronedarone 400mg tablets
  Interventions: Drug: amiodarone

INTERVENTIONS:
Drug: dronedarone (SR33589) — oral administration
  Other Names: Multaq®
  Arms: Dronedarone 400mg bid
Drug: amiodarone — oral administration
  Arms: Amiodarone 600mg/200mg od

SUMMARY:
The objective of this study is to compare the efficacy and safety of dronedarone to that of amiodarone for the treatment of patients with atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented atrial fibrillation for more than 72 hours for whom cardioversion and antiarrhythmic treatment is indicated in the opinion of the investigator and under oral anticoagulation

Exclusion Criteria:

* Contraindication to oral anticoagulation
* Patient having received amiodarone in the past whatever the date (more than a total of twenty 200 mg tablets or more than 5 days intravenous)
* Patients known to have chronic AF, patients with atrial flutter or paroxysmal atrial fibrillation
* Severe congestive heart failure with New-York Heart Association (NYHA) class III or IV, severe bradycardia, high degree atrio-ventricular block, ongoing potentially dangerous symptoms when in AF such as angina pectoris, transient ischemic attacks, stroke, syncope, as judged by the investigator, first degree family history of sudden cardiac death below age 50 years in the absence of coronary heart disease, significant sinus node disease without a permanent pacemaker implanted
* History of torsades de pointes or long QT syndrome or QT- or QTc-interval ≥500 msecs before randomization
* Treatment with other class I or III antiarrhythmic drugs which cannot be discontinued
* Dysthyroidism or other contraindication to amiodarone

The above information are not intended to contain all the considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2007-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: International Clinical Development, Study Director — Sanofi
Locations (23):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Cove, Australia
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Shangaï, China
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Tallinn, Estonia
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Casablanca, Morocco
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Mégrine, Tunisia
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Le Heuzey JY, De Ferrari GM, Radzik D, Santini M, Zhu J, Davy JM. A short-term, randomized, double-blind, parallel-group study to evaluate the efficacy and safety of dronedarone versus amiodarone in patients with persistent atrial fibrillation: the DIONYSOS study. J Cardiovasc Electrophysiol. 2010 Jun 1;21(6):597-605. doi: 10.1111/j.1540-8167.2010.01764.x. Epub 2010 Apr 6. PMID 20384650
- [Derived] Ezekowitz MD. Maintaining sinus rhythm--making treatment better than the disease. N Engl J Med. 2007 Sep 6;357(10):1039-41. doi: 10.1056/NEJMe078148. No abstract available. PMID 17804851

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment of patients started on June 12, 2007 and was completed on October 3, 2008. The study was conducted in 112 centers in 23 countries. Minimum duration of treatment was 6 months. Minimum duration of observation was last patient's randomization plus 190 days.
Pre-assignment Details: Planned sample size was 472. Six hundred and eighteen patients (618) were screened of which 113 did not verify one or more selection criteria. One eligible patient received a placebo capsule (morning intake in the amiodarone group) but was not randomized in the trial. This patient did not report any adverse event and was excluded from all analyses.
Groups:
- Dronedarone 400mg Bid: dronedarone tablets 400mg twice daily (bid)
- Amiodarone 600mg/200mg od: amiodarone 600mg once daily (od) for 28 days, then amiodarone 200mg once daily (od)
Period: Overall Study
Arm/Group | Dronedarone 400mg Bid | Amiodarone 600mg/200mg od
Started | 249 (Randomized and treated patients) | 255 (Randomized and treated patients)
Completed | 153 (completed study drug period) | 186 (completed study drug period)
Not Completed | 96 | 69
Not completed — Lack of Efficacy | 53 | 14
Not completed — Adverse Event | 32 | 45
Not completed — Poor compliance | 6 | 2
Not completed — Not coded/ Not pre-specified | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dronedarone 400mg Bid | Amiodarone 600mg/200mg od | Total
Number analyzed (Participants) | 249 | 255 | 504
Age, Customized [Number; unit: participants]
  18 to < 65 years | 125 | 138 | 263
  65 to < 75 years | 76 | 70 | 146
  >= 75 years | 48 | 47 | 95
Age Continuous [Mean (Standard Deviation); unit: years] | 64.4 (10.8) | 63.7 (10.6) | 64.0 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 73 | 146
  Male | 176 | 182 | 358

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failure
Description: The primary event is the treatment failure defined as the first recurrence of atrial fibrillation or premature study drug discontinuation for intolerance or lack of efficacy according to the investigator judgement. The primary efficacy analysis is performed on the time from first study drug intake to this primary event. The "Measured Values" table below presents the numbers of patients with the event at the end of the study period.
Time Frame: minimum study duration is 6 months (+10 days); maximum is 15 months
Population: All randomized and treated patients (receiving at least one dose of study drug) were included in the efficacy analysis according to the treatment received.
Measure: Number; unit: participants
Arm/Group | Dronedarone 400mg Bid | Amiodarone 600mg/200mg od
Number analyzed (Participants) | 249 | 255
participants | 184 [37.0 to 45.0] | 141 [99.0 to 275.0]
Statistical Analysis 1: Comparison: Dronedarone 400mg Bid vs Amiodarone 600mg/200mg od; Test type: Superiority or Other; p < 0.0001, Log Rank — Cumulative incidence functions in each treatment group were calculated using time-to-event non-parametric Kaplan-Meier estimate. The primary comparison was performed at the 5% level using a 2-sided Log rank test; Hazard Ratio (HR) = 1.59, 95% CI [1.28 to 1.98] — The hazard ratio was estimated by a Cox's proportional hazard model with treatment arm factor. It provides the relative hazard of treatment failure for the dronedarone group compared with the amiodarone group

2. Secondary Outcome: Occurrence of the Main Safety Endpoint (MSE) Defined as Thyroid, Hepatic, Pulmonary, Neurological, Skin, Eye, or Gastrointestinal Specific Treatment Emergent Events or Premature Study Drug Discontinuation Following Any Adverse Event
Description: The considered event is the occurrence of the MSE defined as thyroid, hepatic, pulmonary, neurological, skin, eye, or gastrointestinal specific treatment emergent events or premature study drug discontinuation following any adverse event (AE), whichever comes first. The analysis is performed on the time from first study drug intake to this event. The "Measured Values" table below presents the numbers of patients with the event at the end of the study period.
Time Frame: minimum study duration is 6 months (+10 days); maximum is 15 months
Population: All randomized and treated patients (receiving at least one dose of study drug) were included in the safety analysis according to the treatment received.
Measure: Number; unit: participants
Arm/Group | Dronedarone 400mg Bid | Amiodarone 600mg/200mg od
Number analyzed (Participants) | 249 | 255
participants | 83 | 107
Statistical Analysis 1: Comparison: Dronedarone 400mg Bid vs Amiodarone 600mg/200mg od; Test type: Superiority or Other; p = 0.13, Log Rank — Cumulative incidence functions in each treatment group were calculated using time-to-event non-parametric Kaplan-Meier estimate. The comparison was performed at the 5% level using a 2-sided Log rank test; Hazard Ratio (HR) = 0.80, 95% CI [0.60 to 1.07] — The hazard ratio was estimated by a Cox's proportional hazard model with treatment arm factor. It provides the relative hazard of main safety event occurrence for the dronedarone group compared with the amiodarone group

3. Other Pre Specified Outcome: Occurrence of the MSE Excluding Gastrointestinal Specific Treatment Emergent Events Defined as Diarrhoea, Nausea, Vomiting
Description: The considered event is the occurrence of the MSE excluding gastrointestinal specific treatment emergent events defined as diarrhoea, nausea, vomiting. The analysis is performed on the time from first study drug intake to this event. The "Measured Values" table below presents the numbers of patients with the event at the end of the study period.
Time Frame: minimum study duration is 6 months (+10 days); maximum is 15 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Dronedarone 400mg Bid | Amiodarone 600mg/200mg od
Number analyzed (Participants) | 249 | 255
participants | 61 | 99
Statistical Analysis 1: Comparison: Dronedarone 400mg Bid vs Amiodarone 600mg/200mg od; Test type: Superiority or Other; p = 0.002, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.61, 95% CI [0.44 to 0.84] — The hazard ratio was estimated by a Cox's proportional hazard model with treatment arm factor. It provides the relative hazard of MSE occurrence excluding gastrointestinal events, for the dronedarone group compared with the amiodarone group

ADVERSE EVENTS:
Time Frame: From first to last study drug intake +10 days i.e. end of the study.
Description: The safety population was the "All randomized and treated patients" population.
Arm/Group | Dronedarone 400mg Bid | Amiodarone 600mg/200mg od
Serious Adverse Events (participants affected / at risk) | 34/249 | 37/255
Other Adverse Events (participants affected / at risk) | 146/249 | 165/255
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dronedarone 400mg Bid (N=249) | Amiodarone 600mg/200mg od (N=255)
Cardiac failure (Cardiac disorders) | 6 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 6
Bradycardia (Cardiac disorders) | 1 | 2
Angina pectoris (Cardiac disorders) | 1 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Diastolic dysfunction (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Anaplastic thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoma in situ of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Diverticulitis (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 2
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 | 3
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 2
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 1
Electrocardiogram PR prolongation (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 0 | 2
Death (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0
Mixed liver injury (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Diabetic foot (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Hypoprothrombinaemia (Blood and lymphatic system disorders) | 0 | 1
Symphysiolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dronedarone 400mg Bid (N=249) | Amiodarone 600mg/200mg od (N=255)
Any Gastrointestinal disorders (Gastrointestinal disorders) | 54 | 44
Diarrhoea (Gastrointestinal disorders) | 23 | 8
Nausea (Gastrointestinal disorders) | 13 | 9
Any Infections and infestations (Infections and infestations) | 35 | 35
Any Investigations (Investigations) | 33 | 35
Any Cardiac disorders (Cardiac disorders) | 21 | 36
Bradycardia (Cardiac disorders) | 4 | 14
Any Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 21 | 22
Any Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 21 | 21
Any Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 18 | 23
Any Nervous system disorders (Nervous system disorders) | 17 | 39
Dizziness (Nervous system disorders) | 8 | 16
Any General disorders and administration site conditions (General disorders) | 14 | 26
Oedema peripheral (General disorders) | 6 | 13
Any Vascular disorders (Vascular disorders) | 9 | 23
Hypertension (Vascular disorders) | 7 | 16
Any Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 8 | 17
Any Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 8 | 15
Any Psychiatric disorders (Psychiatric disorders) | 6 | 23
Sleep disorder (Psychiatric disorders) | 3 | 19
Any Eye disorders (Eye disorders) | 6 | 13
Any Endocrine disorders (Endocrine disorders) | 3 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such publication for comment at least 45 days before any submission for publication. If requested by the Sponsor, any submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.